CLINICAL TRIAL: NCT05626842
Title: The 'DR-EAM' Study - (Type 2) Diabetes Weight Reduction - Evaluation of Appcoaching Model
Brief Title: The DR-EAM Type 2 Diabetes Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oviva UK Ltd (Other)
Collaborators: University of Westminster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR-EAM study Oviva; IRAS ID: 269780 (Other: Heath Research Authority (HRA))
Record Dates: First submitted 2022-11-02; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Low calorie diet; Total diet replacement; behaviour change
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): Single-arm real-world evaluation with a matched control group from comparable GP practices
  Interventions: Other: Total Diet Replacement (800kcal/day)

INTERVENTIONS:
Other: Total Diet Replacement (800kcal/day) — The TDR intervention involves a low-calorie, nutritionally complete diet for 12 weeks consuming four meal replacement products exclusively per day, followed by a 4-week food-based reintroduction period; and then weight loss maintenance support monthly for a further 36 weeks. If a patient gains more than 2kg in the maintenance phase, they have the option to follow a TDR for an additional 4 weeks.
  Other Names: TDR; Low energy diet

SUMMARY:
The goal of this 12-month interventional study is to analyse the clinical outcome benefits, scalability and cost-effectiveness of a digital Low-Calorie digital Type 2 diabetes mellitus (T2DM) remission program compared to usual National Health System (NHS) care.

DETAILED DESCRIPTION:
Low-Calorie Diets (LCD) have recently gained popularity as a means of achieving an average 10kg weight loss, 10mmol/mol HbA1c reductions, 50% medication reductions, and Type 2 diabetes mellitus (T2DM) remission (defined as blood-glucose levels <48mmol/mol and off all diabetes-related medications). If these clinical outcomes could be achieved at scale in the United Kingdom, the potential savings for the National Health System (NHS) from reductions in T2DM complications and medication costs are very significant. However, face-to-face T2DM LCD programs are hard to scale due to challenges of accessibility, capacity, and cost.

This single-arm real-world evaluation with a matched control group from comparable GP practices will evaluate clinical outcome benefits and NHS return on investment of a digital LCD program with integrated behavior change intervention.

The 197 will be recruited from GP practices across South West London and Buckinghamshire. Participants will complete a 12-week Total Diet Replacement (TDR) which involves a low-calorie (800kcal/day), nutritionally complete diet, followed by a 4-week food-based reintroduction period; and weight loss maintenance support monthly to 12 months. If a participant gains more than 2kg in the maintenance phase, they have the option to follow a TDR for an additional 4 weeks.

The intervention will be led by Diabetes Specialist Dietitians (DSD) via the Oviva app, telephone, or video calls. All participants will have access to supporting learning materials. Participants will receive intensive support in the first 16 weeks; follow-up support for a further 36 weeks, plus a further 12 months of 'Active follow-up'. Participants finish the trial at 24 months.

After completion, participants continue to receive free access to the Oviva app and their connected monitoring devices.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Maximum age of 65 years
* Male or female
* Minimum BMI of 27kg/m2 (adjusted to 25kg/m² in people of South Asian or Chinese origin)
* BMI <45kg/m2
* T2DM diagnosed at any time
* HbA1c eligibility, most recent value, which must be within 12 months:
* HbA1c ≥ 43 mmol/mol if on diabetes medication
* HbA1c ≥ 48 mmol/mol if on diet alone
* HBA1c <108 mmol/mol
* If HbA1c 90-108 mmol/mol, the value must be within 3 months of referral
* On, or about to start, a second-line diabetes-related medication (metformin is first-line)
* Access to blood glucose monitoring equipment if on a sulphonylurea prior to referral
* Ability to speak, read and receive care in English
* Access to and willing to use an iOS or Android smart phone for the duration of the intervention

Exclusion Criteria:

* T2DM either diet-controlled alone, or on metformin alone
* Current insulin use
* Pregnant or breastfeeding or considering pregnancy during next 6 months
* Significant physical comorbidities:
* Active cancer
* Myocardial infarction or stroke within previous 6 months
* Severe heart failure defined as equivalent to the New York Heart Association grade 3 (NYHA)
* Recent eGFR <30 mls/min/1.73 m2
* Active live disease (except for NAFLD), or a history of hepatoma, or <6 months of onset of acute hepatitis
* Severe angina, cardiac arrythmia including atrial fibrillation or prolonged QT syndrome
* Active substance use disorder / eating disorder
* Porphyria
* Weight loss >5% body weight within last 6 months or on current weight management programme or had/awaiting bariatric surgery (unless willing to come off waiting list)
* Health professional assessment that the person is unable to understand or meet the demands of the treatment programme and/or monitoring requirements, which may include -Learning disabilities
* Taking monoamine-oxidase inhibitor medication
* Taking warfarin
* Taking varenicline (smoking cessation medication)
* Retinopathy diagnosis or lack of retinal screening in the last year
* Active/investigation for gastric or duodenal ulcers
* People currently participating in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary study objective-weight | at baseline, 3, 6, 9,12 & 24 months
  Change in weight (kg) and BMI (kg/m2) continuously via BodyTrace scales
Primary study objective- HbA1c | at baseline, 6, 12 & 24 months
  Change in HbA1c- Diabetes remission defined as 2 HbA1c readings < 48mmol/mol without diabetes medications at least 6 months apart

SECONDARY OUTCOMES:
Secondary study objective- blood pressure | at baseline, 12 & 24 months
  Change in blood pressure (systolic and diastolic) via British and Irish Hypertension Society validated monitors
Secondary study objective- lipids | at baseline, 12 & 24 months
  Change in lipid markers (total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides) via venous sample
Secondary study objective- physical activity | at baseline, 3, 6, 9,12 & 24 months
  continuously via the Fitbit device
Secondary study objective- quality of life | at baseline, 6, 12 & 24 months
  change in quality of life via EQ-5D form
Secondary study objective- participant experience | at 12 months
  via NHS Friends & Family Test standardised survey

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Jones, Study Director
Locations (1):
- Oviva UK ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No